CLINICAL TRIAL: NCT02568579
Title: Effects of Breastfeeding in Immunologic Priming in Young Infants
Brief Title: Infant Immunity Comparison of Breastfed and Bottlefed Infants
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of South Florida (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00050219
Record Dates: First submitted 2015-09-15; First posted 2015-10-06 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2017-06

CONDITIONS: Infant Immunity Response and Immunoglobulin Diversity
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Four 2.6 ml ACD tubes will be collected . All blood will be processed for pyrosequencing, TBNK, CBC and differential, platelets, sera plasman and PBMC's. Stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breastfed: collection of blood/stool/breast milk samples and information about feeding changes and introduction of solid foods. - Cord Blood sample, stool samples monthly and blood sample at 6 month and 12 months of age
  Interventions: Procedure: blood sample/ stool sample
- Bottlefed: collection of blood/stool samples and information about feeding changes and introduction of solid foods. Coord blood sample, stool samples monthly and blood sample at 6 month and 12 month of age.
  Interventions: Procedure: blood sample/ stool sample

INTERVENTIONS:
Procedure: blood sample/ stool sample — blood sample to be done when possible with standard of care lab draw. Stool sample to be collected monthly at home.

SUMMARY:
This study will follow 40 healthy, vaginally delivered infants that are primarily (>/- 75%) breast fed and 40 infants that are exclusively formula fed for at least the first 4 months of life from birth until 12 month age. Visits - Subjects will be consented prior to delivery, visit 1. Subject will be seen if possible after delivery for instruction on stool collection and distribution of supplies, visit 2. Subject will be seen at 6 months of age post immunization, visit 3. Subject will be seen prior to 12 month visit. Study staff will contact via phone/email to collect information about feeding changes.

DETAILED DESCRIPTION:
Cord Blood will be collected at birth if possible and peripheral blood will be collected at 6 month of age (5 to 10 days after receiving their standard 6 month immunizations) and at 12 months of age prior to their 12 month immunization. Additionally, stool samples will be collected within the first week of live and once monthly through 12 months of age. Breastfeeding mothers will collect breast milk once monthly at the same time as the stool specimen during the period of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Self-declared pregnant woman
* Age 18 years or older at the time of consent
* Willing and able to sign consent and follow study schedule
* Planned vaginal delivery
* Willing to primarily breastfed or formula feed for the first four months

Exclusion Criteria:

* Planned delivery by C-Section
* Unwillingness to exclusively breast feed or formula feed their infant for at least the first 4 months
* Unwillingness to receive standard immunizations on the schedule recommended by the American Academy of Pediatrics
* Chronic maternal condition that may influence infant immunity including but not limited to: maternal HIV, immunodeficiency, use of immunosuppressive medications, malignancy or autoimmunity
* Known fetal medical conditions such as congenital malformations
* Use of immune modulating/immune suppressive medication and prophylactic antibiotics during pregnancy
* Any condition that may prevent a mother who plans to breast feed from breast feeding
* Any condition that in the opinion of the investigator would interfere with the conduct of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Pregnant women 18 years of age or older.
  * Vaginal delivery
  * Healthy, full-term babies.
  * Willing to primarily (> 75%) breastfeed or exclusively formula feed for at least the first 4 months of life.
  * Willing to follow the American Academy of Pediatrics' Immunizations guidelines.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Molecular profile of human IgG and IgA by pyrosequencing. | 12 months
  B cell priming and immunoglobulin diversity following immunizations at 2 and 4 month of age by modulating the microbial colonization of infant gut by pyrosequencing by using isotype specific primers.

SECONDARY OUTCOMES:
Vaccine response | 12 months
  post immunization antibody titers (via ELISA) to Hib, tetanus, diphtheria, pertussis and pneumococcal polysaccharide serotypes contained in the Prevnar 13 vaccine.
Antibody activity | 12 months
  Functional activity of antibodies measured by opsonophagocytic activity to Pneumococcal and Hib vaccine
Plasma level of B cell activating factor and/or a proliferation-inducing ligand | 12 months
  Degree of B cell differentiation and activation in B cell by BD bioscience Canto flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: John Sleasman, MD, Study Director — Duke University
Locations (3):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina